CLINICAL TRIAL: NCT06431945
Title: Early Detection of Hepatitis C in Injection Drug Users
Brief Title: Early Detection of HCV in Injection Drug Users
Acronym: EDVIP
Status: Recruiting | Type: Observational
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: Institute for Clinical and Experimental Medicine (Other Government); Brno University Hospital (Other); České Budějovice Hospital (Other); University Hospital Hradec Kralove (Other); University Hospital Olomouc (Other); Hepatogastroenterology Hradec Kralove (Unknown); Regional Hospital Karlovy Vary (Unknown); Clinic Podane ruce (Unknown); Tomáš Baťa Regional Hospital in Zlín (Unknown); Hospital Agel Prostějov (Unknown); Hospital Jihlava (Unknown); Hospital Havířov (Unknown); Hospital Tábor (Unknown); Remedis Prague (Unknown); Hospital Opava (Unknown); Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other); Military University Hospital, Prague (Other); Hospital Pardubice (Unknown)
Responsible Party: Sponsor
Other Study IDs: UZIS 2023/1
Record Dates: First submitted 2024-04-23; First posted 2024-05-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV; PWID; Point of care testing; Hepatitis; Czech Republic; HCV genotype
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People who inject drugs
  Interventions: Diagnostic Test: Hepatitis C antibody (anti-HCV) test; Diagnostic Test: Hepatitis C RNA test and genotype test

INTERVENTIONS:
Diagnostic Test: Hepatitis C antibody (anti-HCV) test — Testing for hepatitis C antibodies determines whether or not you have been exposed to HCV at some point in your life. This testing will be performed in all 3,000 persons who inject drugs enrolled in the project.
Diagnostic Test: Hepatitis C RNA test and genotype test — RNA is a type of genetic material from HCV that can be detected in the blood. This test will be used as a confirmation of the infection. This testing will be performed in all persons with positive antibody test who will come to clinical center.

SUMMARY:
The project is a national, prospective, multicenter, non-interventional pilot project of screening HCV in PWID in the Czech Republic.

The main goal of the project is to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure of early detection of Hepatitis C and setting up and testing new methods and implementation into the system of social health care.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, non-interventional pilot project of screening HCV in PWID in 18 clinical centers in the Czech Republic.

The main goal of the project is the elimination of further transmission of hepatitis C virus and to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure of early detection of Hepatitis C and setting up and testing new methods and implementation into the system of social health care.

The project will include testing the procedure on a sample of approx. 3,000 PWID which can help to identify weak points in the continuum of care. A methodology for the continuous care of the target group in the early diagnostic and therapeutic stages will be created. Proposal for a system change towards streamlining the screening process.

The project is supported by the European Social Fund (Operational Program Employment plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0000281.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* an active injecting drug user or have used injecting drugs at any time in the past

Exclusion Criteria:

* not agreeing to participate in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any people who inject drugs with age 18+ tested by cetres participating in the project.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of the hepatitis C virus in screened cohort of persons who inject drugs | Until 31. 12. 2025

SECONDARY OUTCOMES:
Up to 3,000 persons who inject drugs (PWID) enrolled in the project | Until 31. 12. 2025
Optimal methodological settings for early detection of the Hepatitis C virus based on hepatitis C antibody and hepatitis C RNA testing | Until 31. 12. 2025

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Mravcik, assoc. prof., Study Director — Charles University First Faculty of Medicine
Locations (18):
- Czechia (18):
  - Brno University Hospital, Brno
  - Clinic Podane ruce, Brno
  - České Budějovice Hospital, České Budějovice
  - Hospital Havířov, Havířov
  - Hepatogastroenterology Hradec Kralove, Hradec Králové
  - University Hospital Hradec Kralove, Hradec Králové
  - Hospital Jihlava, Jihlava
  - Regional Hospital Karlovy Vary, Karlovy Vary
  - University Hospital Olomouc, Olomouc
  - Hospital Opava, Opava
  - Hospital Pardubice, Pardubice
  - Institute for Clinical and Experimental Medicine, Prague
  - Military University Hospital, Prague, Prague
  - Remedis Prague, Prague
  - Hospital Agel Prostějov, Prostějov
  - Hospital Tábor, Tábor
  - Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s., Ústí nad Labem
  - Tomáš Baťa Regional Hospital in Zlín, Zlín

IPD SHARING:
Plan to Share IPD: No